CLINICAL TRIAL: NCT06841302
Title: Investigation of Alexithymia Levels in Fibromyalgia Syndrome Before and After Treatment
Brief Title: Alexithymia Levels in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, MD, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstPRMTRH-EK
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia (FM); Alexithymia
Keywords: Fibromyalgia; Alexithymia; aerobic exercise
MeSH Terms: conditions — Fibromyalgia; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Fibromyalgia (Experimental): This study group consisted of individuals diagnosed with fibromyalgia syndrome (FMS) according to the American College of Rheumatology criteria, who were also literate. The study specifically excluded individuals with pre-existing psychiatric disorders, neurological conditions known to cause alexithymia, or those currently undergoing antidepressant treatment. All study participants were enrolled in a combined treatment program consisting of both a structured aerobic exercise program (swimming, cycling, or brisk walking for at least three days a week, with each session lasting two hours) and a pharmacological treatment regimen. Patients who did not adhere to the prescribed treatment regimen or who discontinued follow-up were excluded from the study.
  Interventions: Other: Fibromyalgia Agents

INTERVENTIONS:
Other: Fibromyalgia Agents — All study participants were enrolled in a combined treatment program consisting of both a structured aerobic exercise program (swimming, cycling, or brisk walking for at least three days a week, with each session lasting two hours) and a pharmacological treatment regimen. Patients who did not adhere to the prescribed treatment regimen or who discontinued follow-up were excluded from the study.

SUMMARY:
The primary aim of this study was to investigate the changes in alexithymia levels in fibromyalgia patients over a six-month period following a combined treatment and to assess the relationship between changes in fibromyalgia symptom severity and changes in alexithymia levels. Specifically, the study sought to determine if improvements in fibromyalgia symptoms, as measured by the Visual Analog Scale (VAS), were associated with reductions in alexithymia, as measured by the Toronto Alexithymia Scale-20 (TAS-20).

DETAILED DESCRIPTION:
Background and Objectives: Fibromyalgia (FM) is a chronic pain condition characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and cognitive difficulties. FM affects approximately 0.2-6.6% of the world's population and is more frequent in women. It is known that psychiatric comorbidities are frequently observed in individuals with fibromyalgia (FM). In this context, while depression/major depressive disorder (MDD) stands out as the most commonly encountered psychiatric disorder among individuals diagnosed with FM, bipolar disorder, panic disorder, post-traumatic stress disorder (PTSD), and less frequently, anxiety disorders are also observed. The presence of these comorbidities can affect the clinical course and treatment response of FM, therefore, it is important to consider this condition in the evaluation of FM patients and in the development of treatment plans.

Alexithymia, characterized by difficulty identifying and describing feelings and a preference for external thinking, potentially leading individuals to report somatic symptoms like pain rather than emotional experiences. Alexithymia is more prevalent in individuals with fibromyalgia and it correlates with both distress and pain intensity. This study investigates whether successful SSRI treatment in fibromyalgia patients correlates with improved alexithymia levels, exploring the potential link between treatment response and enhanced emotional processing.

Methods:This prospective observational cohort study was conducted at Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. Patients diagnosed with fibromyalgia syndrome (FMS) according to American College of Rheumatology criteria were included. Those with psychiatric disorders, neurological conditions causing alexithymia, or under antidepressant treatment were excluded. All participants received duloxetine treatment combined with an aerobic exercise program. Fibromyalgia symptoms were assessed using Visual Analog Scale (VAS) at baseline and 6 months, while alexithymia was evaluated using Toronto Alexithymia Scale-20 (TAS) at baseline, 3, and 6 months. Statistical analysis included repeated measures ANOVA with Greenhouse-Geisser correction, paired t-tests, and correlation analyses, with adjustments for age, BMI, and daily medication count.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology's Fibromyalgia diagnostic criteria Have not received any previous psychiatric treatment

Exclusion Criteria:

* Presence of psychiatric disorders History of antidepressant use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Alexithymia Level | From enrollment to the end of treatment at 6 months
  The primary outcomes of this study are changes in alexithymia levels, measured by the Toronto Alexithymia Scale-20 (TAS-20), over the six-month period of treatment follow up.
VAS score | From enrollment to the end of treatment at 6 months
  Changes in participants' fibromyalgia symptom severity were measured with a Visual Analog Scale (VAS).
Correlations between baseline values and post-treatment changes | From enrollment to the end of treatment at 6 months
  The examination of associations between baseline Toronto Alexithymia Scale and Visual Analog Scale scores and posttreatment changes in these measures to investigate whether baseline symptom severity or alexithymia levels were predictive of treatment response.

SECONDARY OUTCOMES:
Changes in TAS subscales | From enrollment to the end of treatment at 6 months
  Changes in the individual subscales (e.g., Difficulty Identifying Feelings, Difficulty Describing Feelings, Externally-Oriented Thinking) could be considered secondary outcomes, providing a more granular understanding of how alexithymia is affected.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Physical Medicine and Rehabilitation Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Martinez MP, Sanchez AI, Miro E, Lami MJ, Prados G, Morales A. Relationships between physical symptoms, emotional distress, and pain appraisal in fibromyalgia: the moderator effect of alexithymia. J Psychol. 2015 Jan-Apr;149(1-2):115-40. doi: 10.1080/00223980.2013.844673. Epub 2014 Mar 5. PMID 25511201
- [Background] Sfarlea A, Dehning S, Keller LK, Schulte-Korne G. Alexithymia predicts maladaptive but not adaptive emotion regulation strategies in adolescent girls with anorexia nervosa or depression. J Eat Disord. 2019 Nov 29;7:41. doi: 10.1186/s40337-019-0271-1. eCollection 2019. PMID 31798880
- [Background] Di Tella M, Castelli L. Alexithymia and fibromyalgia: clinical evidence. Front Psychol. 2013 Dec 2;4:909. doi: 10.3389/fpsyg.2013.00909. eCollection 2013. PMID 24348453
- [Background] Kleykamp BA, Ferguson MC, McNicol E, Bixho I, Arnold LM, Edwards RR, Fillingim R, Grol-Prokopczyk H, Turk DC, Dworkin RH. The Prevalence of Psychiatric and Chronic Pain Comorbidities in Fibromyalgia: an ACTTION systematic review. Semin Arthritis Rheum. 2021 Feb;51(1):166-174. doi: 10.1016/j.semarthrit.2020.10.006. Epub 2020 Dec 29. PMID 33383293
- [Background] Habibi Asgarabad M, Salehi Yegaei P, Jafari F, Azami-Aghdash S, Lumley MA. The relationship of alexithymia to pain and other symptoms in fibromyalgia: A systematic review and meta-analysis. Eur J Pain. 2023 Mar;27(3):321-337. doi: 10.1002/ejp.2064. Epub 2022 Dec 20. PMID 36471652
- [Derived] Atasoy M, Kalaoglu E, Takim U, Gokcay H. Investigation of alexithymia levels in fibromyalgia before and after treatment. Clin Exp Rheumatol. 2026 Jan;44(1):130-137. doi: 10.55563/clinexprheumatol/45nmy7. Epub 2025 Oct 3. PMID 41042725